CLINICAL TRIAL: NCT07390136
Title: SPRINT: Sparking Potential, Revealing Infant Neurocognitive Traits
Brief Title: Sparking Potential, Revealing Infant Neurocognitive Traits
Acronym: SPRINT
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0452; UWMSN | SMPH | NRL Neurology (Other: UW Madison); Protocol Version 5/3/2024 (Other: UW Madison)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Perinatal Brain Injury; Healthy Participants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with perinatal brain injuries: Children ages 6 months (may be enrolled prior to 6 months) - 24 months who are diagnosed with 1) hypoxic- ischemic encephalopathy, 2) cerebral palsy, and/or 3) were born premature at less than 28 weeks gestational age.
- Healthy Children: Children ages 6 months (may be enrolled prior to 6 months) - 24 months of age with no prior history of a brain and/or cardiac illness early in life.

SUMMARY:
This research focuses on the long-term cognitive development of children, including healthy infants and those who had a perinatal brain injury. As part of this research study, children complete virtual game and assessments. Parents will be asked to fill out questionnaires about their child's behavior and stress in the home. All study visits will take place online via Zoom.

ELIGIBILITY:
Inclusion Criteria:

* Child-parent dyads will be recruited to the study.
* Children 3-24 months with and without a history of a perinatal brain injury (PBI) will be included in this study.
* Children with PBIs will include:

  * Children diagnosed during the neonatal period with hypoxic-ischemic encephalopathy,
  * Children born at a premature gestational age (born at less than 32 weeks gestational age).
  * Children diagnosed with cerebral palsy
* Healthy control participants meeting inclusion criteria will include:

  * healthy infants with no prior neurological (brain disorder) history
* For all parents: the only research inclusion criteria is to be the parent or legal guardian of a newborn with perinatal brain injury or healthy control participant.

Exclusion Criteria:

* Healthy infants to be included in the control group will not have:

  * a prior history of brain injury
  * a diagnosis of cerebral palsy
  * a history of a neurological disorder
  * prior admission to the Neonatal Intensive Care Unit (NICU)
* Children with chromosomal abnormalities, genetic syndromes and major congenital malformations will be excluded from both the patient groups and the control group.
* Parents will have no exclusionary criteria.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants ages 6-24 months located across the United States and internationally.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Infant Attention Task (IAT) | Assessed at the 12,18, and 24-month time points
  A behavioral measure used with infants to assess attentional control and processing. Infants are presented with visual puppet stimuli four distinct "looks", and researchers record looking time, shifts in attention, or habituation patterns. More sustained attention in the early looks followed by habituation to the stimuli in the later looks often indicates better early attentional capacity. Total accumulated looking time to a stimulus in visual preference-type tasks commonly ranges from roughly 15-30+ seconds per trial, depending on the infant's age and the stimulus.
Cognitive Adaptive Test/Clinical Linguistic & Auditory Milestone Scale (CAPUTE) | Assessed at the 6 and 12-month time points
  An assessment for infants and young children that evaluates cognitive and language development. It combines two scales: CAT (Cognitive Adaptive Test) for problem-solving and adaptive skills, and CLAMS (Clinical Linguistic and Auditory Milestone Scale) for language and auditory milestones. Scores provide age-equivalent estimates of cognitive and language abilities. The CAPUTE scores are reported as developmental quotients ranging roughly from 40 to 160, with scores ≥85 considered within normal limits, 70-84 indicating borderline development, and <70 suggesting developmental delay.

SECONDARY OUTCOMES:
Confusion, Hubbub and Order Scale (CHAOS) | Assessed at the 6, 9,12, and 24-month time point
  Parents and/or Caregivers rate items describing household noise, crowding, and routine; responses are summed to create a total CHAOS score. The CHAOS total score ranges from 15 to 60, with higher scores indicating a more chaotic, noisy, and disorganized home environment; scores below 25 typically reflect lower chaos, whereas scores above 35 suggest high household chaos.
Parental Stress Scale | Assessed at the 6,12,18, and 24-month time points
  A questionnaire which measures stress and satisfaction associated with parenting; items are summed to create a total parental stress score. On the Parental Stress Scale, total scores range from 18 to 90, with higher scores indicating greater levels of parental stress and lower scores reflecting lower stress and more satisfaction in the parenting role.
Parenting Daily Hassle (PDH) Scales: Frequency Score | Assessed at the 6,12,18, and 24-month time point
  A parent-report measure assessing the frequency and intensity of everyday parenting stressors (e.g., child demands, disruptions to routines); item ratings are summed or averaged to yield frequency and intensity scores. On the PDH Scale, frequency scores range from 0 to 80 with higher totals indicating more frequent and/or more stressful everyday parenting hassles.
Parenting Daily Hassle (PDH) Scales: Intensity Score | Assessed at the 6,12,18, and 24-month time point
  A parent-report measure assessing the frequency and intensity of everyday parenting stressors (e.g., child demands, disruptions to routines); item ratings are summed or averaged to yield frequency and intensity scores. On the PDH Scale, intensity scores range from 0 to 100 with higher totals indicating more frequent and/or more stressful everyday parenting hassles.
Pediatric Quality of Life Inventory (Peds-QL) | Assessed at the 6, 9,18, and 24-month time point
  The PedsQL is an inventory of statements scored by reverse-scoring responses to a 5-point Likert scale and then transforming them to a 0-100 scale. A higher score indicates a better quality of life.
Early Executive Function Questionnaire (EEFQ) | Assessed at the 6, 9,18, and 24-month time points
  A questionnaire is given to parents that assesses what executive functions children are exhibiting. More functions exhibited means further along in executive function development. The (EEFQ uses parent ratings on a 7-point scale for 31 items, with subscale and composite scores averaging between 1 and 7 - higher scores indicate stronger emerging executive function behaviors in infants and toddlers.
Reilly Role Overload Questionnaire | Assessed at the 6, 9,18, and 24-month time point
  In the Reilly Role Overload questionnaire, parents of child participants rate the frequency of feeling overwhelmed by role demands; item responses are summed to create a total role overload score. Total scores range from 13 to 65, with higher scores indicating greater perceived role overload due to excessive demands relative to time and energy.
Behavior Rating Inventory of Executive Function-Preschool (BRIEF-P) | Assessed at the 24-month time point
  Behavior is reported in the BRIEF-P. Behaviors reported by parents can be used to predict later executive function exhibited by children. List of statements provided about child's behavior, parent will answer whether this is never a problem (N), sometimes a problem (S), and often a problem (O). Responses reported as participant counts, answering N more often is considered a better score. On the BRIEF-P, T-scores around 50 are average, 60-64 are slightly at risk, and 65 or higher indicate significant executive function difficulties.
Parent Report of Children's Abilities-Revised (PARCA-R) | Assessed at the 24-month time point
  The PARCA-R is a parent-completed questionnaire used to assess early cognitive and language development in young children (around 2 years old). It asks parents about their child's vocabulary, sentence use, and nonverbal skills. Parents' responses are summed to generate language, nonverbal, and total cognitive scores. Scores have a mean of 100, with scores around 100 indicating typical cognitive and language development at approx. 2 years, lower scores suggesting possible delay, and higher scores reflecting stronger development

CONTACTS AND LOCATIONS:
Overall Officials: Melisa Carrasco McCaul, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuevas K, Bell MA. Infant attention and early childhood executive function. Child Dev. 2014 Mar-Apr;85(2):397-404. doi: 10.1111/cdev.12126. Epub 2013 May 24. PMID 23711103